CLINICAL TRIAL: NCT05709340
Title: Efficacy of PNF Exercises on Treatment of Temporomandibular Dysfunction in Patients With Forward Head Posture: A Double-blind, Randomized, Controlled Trial
Brief Title: PNF Exercises on Treatment of Temporomandibular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNF exercises for TMJ
Record Dates: First submitted 2023-01-21; First posted 2023-02-02 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: proprioceptive neuromuscular facilitation exercises
- control group (Active Comparator)
  Interventions: Other: traditional physical therapy treatment

INTERVENTIONS:
Other: proprioceptive neuromuscular facilitation exercises — PNF exercises will be done for Masseter, Temporalis, Lateral pterygoid and medial pterygoid muscles. Each contraction will be held for 10 seconds, and each stretch (relaxation phase) will be allowed to continue as long as the muscle tension continued to give away.
  Arms: study group
Other: traditional physical therapy treatment — * Ultrasound: Continuous ultrasound at 1MHZ to temporomandibular joint at 1.0-1.25 W/CM2 for 5 min over each affected TMJ and masseter area, with the mouth in a slightly open position.
  * Forward head posture correction exercises including: chin tuck exercise, Strengthening shoulder retractors, stretching of sternocleidomastoid muscle, and Stretching of pectoralis muscle.
  Arms: control group

SUMMARY:
Temporomandibular joint dysfunction (TMJD) is an important health problem that occurs approximately in 22 to 35 percent of adults, different physiotherapy methods are reported as treatment options for management of TMJD. Although that, there is no previous studies about the efficacy of PNF exercises in treatment of TMJD in patients with forward head posture. So, the purpose of the present double-blind, randomized, controlled trial is to investigate the efficacy of PNF exercises in treatment of TMJD in patients with forward head posture.

ELIGIBILITY:
Inclusion criteria:

* Patients of both genders of age between 20-40 years
* having symptoms of TMD for at least six weeks duration established by an expert physician or orthopaedician
* having forward head posture with CVA < 53
* pain over TMJ between 3 to 6 on NPRS
* mouth opening < 25mm.

Exclusion criteria:

Patients will be excluded if they exhibited any of the following criteria:

* TMJ fracture undergone any surgical procedure for TMJ
* Fracture surrounding TMJ
* Dislocation or subluxation of TMJ
* systemic generalized joint diseases, such as rheumatoid arthritis, and osteoporosis, congenital diseases, or facial paralysis
* recently any dental treatment is taken or surgery over TMJ
* hematological cervical disorders which may affect the jaw
* Neurological deficits e.g. Bells palsy, Trigeminal neuralgia.
* Recent infections (within the last six months) affecting the head and neck e.g. bone infections, meningitis, encephalitis, malaria, ear infection
* Participants who were using any functional appliances e.g. dentures, braces, bite appliances which had been adjusted or fitted in the last 12 weeks prior to the commencement of this study
* DDwR, DDwoR
* Patients were excluded from the study if they were receiving any other form of treatment for their TMJ dysfunction.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | change from base line at 6 weeks.
  A pressure algometer will be used for the objective measurement of the PPT. The algometer was pressed on the masseter, temporalis muscles until the patient feel pain. The unit of measurement will be in kg/cm2, and three measurements will be taken every 30 seconds. The average of the three consecutive measurements will be taken as the final value.

SECONDARY OUTCOMES:
ROM assessment | change from base line at 6 weeks.
  A caliper will be used to measure mandibular depression, protrusion and lateral deviation.
Temporomandibular Disorder Disability Questionnaire | change from base line at 6 weeks.
  This questionnaire consists of the following:
  * The Temporomandibular Disorder Disability Index. It consists of 10 questions with 5 possible answers, rating a 0 to 4 score level for each of the answers.
  * The Temporomandibular Disorder symptom intensity scale and the Temporomandibular Disorder symptom frequency scale are two visual analogue scales which address the frequency and intensity of a patient's TMJ symptoms and consist of 7 sections for each scale where the patient must rate his/her intensity and frequency of symptoms on a scale of 0 to 10 score level.
  * The Pain Drawing sheet is used by the patients to capture pain location and quality.
Numerical Rating Scale (NRS) | change from baseline at 6 weeks.
  The patient will be asked to indicate a number between 0 and 100 on a horizontal line, that best described his/her perceived level of pain intensity when it is at its worst and when it is at is least. The average of these two totals indicates the average pain experienced by the patient as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- marwa S saleh, Giza, Egypt